CLINICAL TRIAL: NCT07291986
Title: Comparing Visual Outcomes After FemtoLasik and Implantable Collamer Lens in Treatment of Myopia
Brief Title: To Compare the Clinical Outcomes of FemtoLASIK and ICL Implantation in Treating Moderate Myopia Focusing on Refractive Stability, Contrast Sensitivity and High Order Aberrations.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walid Osama Abdel Rahman Nour El Din (Other)
Responsible Party: Sponsor-Investigator, Walid Osama Abdel Rahman Nour El Din, Cornea and Refractive Ophthalmology Consultant, Fayoum University
Organization: Fayoum University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D261
Record Dates: First submitted 2025-11-25; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Myopia, Moderate
Keywords: FemtoLASIK, ICL, myopia, HOA, contrast sensitivity
MeSH Terms: conditions — Myopia; Lymphoma, Follicular; T-Lymphocytopenia, Idiopathic CD4-Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simple Myopic Patients (Active Comparator): Patients with simple myopia undergoing FemtoLASIK or ICL surgeries
  Interventions: Procedure: FemtoLASIK; Procedure: ICL implantation
- Compound Myopic Patients (Active Comparator): Patients with compound myopia undergoing FemtoLASIK or ICL surgeries
  Interventions: Procedure: FemtoLASIK; Procedure: ICL implantation

INTERVENTIONS:
Procedure: FemtoLASIK — FemtoLASIK surgery for simple and compound myopic patients
Procedure: ICL implantation — ICL implantation for simple and compound myopic patients

SUMMARY:
Compare the clinical outcomes of FemtoLASIK and ICL implantation in treating moderate myopia.

DETAILED DESCRIPTION:
The clinical outcomes of FemtoLASIK and ICL implantation focusing on refractive stability, contrast sensitivity and high order aberrations.

ELIGIBILITY:
Inclusion Criteria:

Group I - FemtoLASIK subgroup:

* Age range: 21-40 years.
* Stable myopia for at least one year (refractive change

  ≤ 0.50 D).
* Spherical equivalent between -4.00 D and -8.00 D.
* Corneal thickness ≥ 500 μm, residual stromal bed > 300 μm and percentage of tissue altered < 39%.
* No evidence of keratoconus or ectatic changes on corneal topography/tomography.
* Mesopic pupil diameter ≤ 6.5 mm.
* Absence of ocular surface disease or significant dry eye symptoms.
* No history of prior ocular surgery or trauma.

Group II - ICL subgroup:

* Age range: 21-40 years.
* Stable myopia (with or without astigmatism) for ≥1 year.
* Spherical equivalent between -4.00 D and -8.00 D.
* Anterior chamber depth ≥ 2.8 mm from endothelium.
* Endothelial cell density ≥ 2500 cells/mm².
* White-to-white and sulcus-to-sulcus diameters suitable for ICL sizing.
* Clear crystalline lens with no signs of early cataract.
* No history of intraocular surgery, uveitis, or glaucoma.

Exclusion Criteria:

Patients with mild myopia (<-4D) or high myopia (>- 8D) or hyperopia.

* Patients with media opacity.
* Patients with associated ocular pathology.
* Patients with corneal topography not fitting to either treatment modalities.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-05-06 (Actual)

PRIMARY OUTCOMES:
Refractive Stability (%) | From enrollment up to 6 months postoperative
  calculating the ratio between spherical equivalent postoperative to that of preoperative
Contrast Sensitivity (log CS) | From enrollment up to 6 months postoperative
  using specialized charts and measured in logarithmic contrast sensitivity (log CS) units
High Order Aberrations (μm) | From enrollment up to 6 months postoperative
  using the RMS value to quantify the total magnitude of wavefront deviations in the eye in micrometers

CONTACTS AND LOCATIONS:
Overall Officials: Omar M Said, MD, Study Director — Faculty of Medicine, Fayoum University
Locations (1):
- Faculty of Medicine, Fayoum University, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT07291986/Prot_SAP_000.pdf